CLINICAL TRIAL: NCT06896357
Title: Effectiveness and Safety of Limbal Relaxing Incisions for Correcting Post Phacoemulsification High Astigmatism
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Youstina shaheir shawky gad, resident doctor of ophthalmology, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LRIs in high astigmatism
Record Dates: First submitted 2025-03-17; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Astigmatism; Phacoemulsification
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients with post phacoemulsification high astigmatism . (Experimental)
  Interventions: Procedure: Limbal relaxing incisions

INTERVENTIONS:
Procedure: Limbal relaxing incisions — A fixed depth diamond-guarded knife (Gemcision LRI 600 Microns Blade, Katalyst Surgical, chesterfield, MO, USA) will be used to create a paired circumferential corneal incision, following the limbal curvature, 1-1.5mm anterior to the limbus centered on the steep corneal meridian. The incision arc length will be ninety degree according to the Nichamin Age and Pachymetry Adjusted (NAPA) nomogram.

SUMMARY:
To compare the effect of Limbal relaxing incisions (LRIs) plus spectacle correction versus spectacle correction alone on subjective and objective improvement in visual function for correcting post phacoemulsification high astigmatism .

DETAILED DESCRIPTION:
Astigmatism is one of the commonest refractive errors encountered during our clinical practice. Surgically induced astigmatism is the main obstacle to achieve good uncorrected visual acuity following cataract surgery. It is estimated that corneal astigmatism of more than 1.0 diopter (D) is found in up to 40% of patients presenting for cataract surgery, 1.5D or more is present in over 20% and above 2.0D in 10%.

Astigmatism induces distortion of the image leading to compromise quality of vision. In order to achieve better visual results, the effect of postoperative astigmatism should be minimized, management options for corneal astigmatism include glasses, contact lenses, and surgery such as Limbal relaxing incisions (LRIs), refractive laser surgery, toric lenses or rarely corneal grafting. The LRIs technique involves the placement of incisions corresponding to the steep meridian, resulting in corneal flattening and the reduction of astigmatic power. LRI is a safe and an inexpensive procedure, which is simple for experts to perform. Although most of the nomograms recommended that LRIs technique can correct up to 3 D of astigmatism ,it has been found that it is possible to correct even more than 4 D if the incisions were performed on high degrees of astigmatism.

ELIGIBILITY:
Inclusion Criteria:

* Conventional phacoemulsification was done at least one month earlier.
* Clear cornea with corneal astigmatism more than 3.0 D.

Exclusion Criteria:

* History of corneal surgeries (e.g., keratoplasty, refractive surgery, and corneal wound repair).
* Ocular trauma.
* Other intraocular surgery.
* Patient with corneal opacities.
* Thin cornea .
* Any significant ocular disease causing diminution of vision (e.g., optic atrophy, diabetic retinopathy, and age-related macular degeneration), autoimmune disease, and peripheral corneal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
visual acuity improvement | 3 months
  assessment the improvement in visual acuity ,which will be measured by Landolt Cs chart with decimal notation.
contrast sensitivity improvement | 3 months
  Assessment the improvement in contrast sensitivity using Pelli-Robson contrast sensitivity test .

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Ismail Ahmed, Professor, Study Chair — Assiut University; Hani Omar Elsodafy, Assistant Professor, Study Chair — Assiut University; Sara Hussein Mohamed, Lecturer, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Li Z, Han Y, Hu B, Du H, Hao G, Chen X. Effect of Limbal relaxing incisions during implantable collamer lens surgery. BMC Ophthalmol. 2017 May 8;17(1):63. doi: 10.1186/s12886-017-0458-7. PMID 28482825
- [Background] Rashwan A, Natag A, Wasfi E, Lotfy H, Shehata MJDJoO. Manually performed limbal relaxing incisions versus femtosecond laser-guided astigmatic keratotomy for correction of corneal astigmatism after phacoemulsification. 2024;25(3):150-5
- [Background] OAM SWJUJoO. Managing Corneal Astigmatism. 2023;11(03):78-82
- [Background] Khan MI, Muhtaseb M. Prevalence of corneal astigmatism in patients having routine cataract surgery at a teaching hospital in the United Kingdom. J Cataract Refract Surg. 2011 Oct;37(10):1751-5. doi: 10.1016/j.jcrs.2011.04.026. Epub 2011 Aug 12. PMID 21840163
- [Background] Ferrer-Blasco T, Montes-Mico R, Peixoto-de-Matos SC, Gonzalez-Meijome JM, Cervino A. Prevalence of corneal astigmatism before cataract surgery. J Cataract Refract Surg. 2009 Jan;35(1):70-5. doi: 10.1016/j.jcrs.2008.09.027. PMID 19101427
- [Background] Theiss MB, Santhiago MR, Moraes HV Jr, Gomes BF. Prevalence of corneal astigmatism in cataract surgery candidates at a public hospital in Brazil. Arq Bras Oftalmol. 2019 Jun 3;82(5):377-380. doi: 10.5935/0004-2749.20190071. PMID 31166427
- [Background] Khoramnia R, Auffarth G, Labuz G, Pettit G, Suryakumar R. Refractive Outcomes after Cataract Surgery. Diagnostics (Basel). 2022 Jan 19;12(2):243. doi: 10.3390/diagnostics12020243. PMID 35204334